CLINICAL TRIAL: NCT03081845
Title: Comparative Effects of A1 Versus A2® Milk on the Gastrointestinal Physiology, Symptoms and Cognitive Behaviour for the Preschool Children: a Double-blinded Randomized Controlled Cross-over Study
Brief Title: A1 Versus A2® Milk on the Gastrointestinal Physiology, Symptoms and Cognitive Behaviour for the Preschool Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: a2 Milk Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 15-SC-5-A2-002
Record Dates: First submitted 2017-02-28; First posted 2017-03-16 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Gut Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A1-A2 (Experimental): Oral consumption of milk A1 in study phase 1. Oral consumption of milk A2 in study phase 2.
  Interventions: Dietary Supplement: Oral consumption of milk A1 in study phase 1; Dietary Supplement: Oral consumption of milk A2 in study phase 2
- Sequence A2-A1 (Experimental): Oral consumption of milk A2 in study phase 1. Oral consumption of milk A1 in study phase 2.
  Interventions: Dietary Supplement: Oral consumption of milk A2 in study phase 1; Dietary Supplement: Oral consumption of milk A1 in study phase 2

INTERVENTIONS:
Dietary Supplement: Oral consumption of milk A1 in study phase 1 — Oral consumption of 250 ml of milk containing both A1 and A2 type beta casein 2 times per day after meal for 5 days in study phase 1.
  Arms: Sequence A1-A2
Dietary Supplement: Oral consumption of milk A2 in study phase 1 — Oral consumption of 250 ml of milk containing only A2 type beta casein 2 times per day after meal for 5 days in study phase 1.
  Arms: Sequence A2-A1
Dietary Supplement: Oral consumption of milk A1 in study phase 2 — Oral consumption of 250 ml of milk containing both A1 and A2 type beta casein 2 times per day after meal for 5 days in study phase 2.
  Arms: Sequence A2-A1
Dietary Supplement: Oral consumption of milk A2 in study phase 2 — Oral consumption of 250 ml of milk containing only A2 type beta casein 2 times per day after meal for 5 days in study phase 2.
  Arms: Sequence A1-A2

SUMMARY:
This is a multiple-sites, double-blinded, randomized, controlled, parallel-designed, cross-over study among healthy preschoolers with 5 days consumption of A2 or A1 milk to compare the effects on gut inflammation, gastrointestinal symptoms and behavioral well-being.

DETAILED DESCRIPTION:
Gut inflammation is reflected by serum C-Reactive Protein (CRP), hemoglobin (HB), interleukin-4 (IL-4), Immunoglobulin G (IgG), Immunoglobulin E (IgE), Immunoglobulin G1 (IgG1), Immunoglobulin G2a (IgG2a), β-Casomorphin-7 (BCM-7), Glutathione, calcium (Ca), iron (Fe) and zinc (Zn) concentration; gastrointestinal (GI) symptoms are measured via Visual Analog Scale (VAS) for gut tolerance, including borborygmus, bloating, break wind, abdominal pain, and diarrhea; behavioral well-being is assessed using Subtle Cognitive Impairment Test (SCIT).

The total duration of study was 24 weeks, including subject enrollment, study intervention, laboratory testing, and providing clinical study report. The cross-over study consisted of 5 days of each product intervention; 10 days of wash-out in phase 1 and phase 2, respectively; and then followed by 6 weeks of statistical analysis and clinical report completion.

ELIGIBILITY:
Inclusion Criteria:

* Non-regular milk drinker;
* Suffered from mild to moderate milk intolerance;
* Agree not to take any medication, supplements, nutrition or other dairy products including acidophilus milk;
* Parent(s) or legal guardian's consent to the study and willing to comply with study procedures;
* Parent(s) or guardian of infant agrees not to enroll infant another clinical study while participating in this study;
* Fully understand the nature, objective, benefit and the potential risks and side effects of the study.

Exclusion Criteria:

* Have known dairy allergy;
* Suffered from severe milk intolerance;
* Unable to give written informed consent;
* Use of antibiotics at the time of screening, or during the past two weeks;
* Have history of fecal impaction;
* Trying to lose weight by following a diet or exercise regimen designed for weight loss, or taking any drug influencing appetite and any drug for weight loss for the last three months;
* Have participated in similar dairy or probiotics-containing product's clinical trials within 3 months before the screening;
* Currently taking medicines for cardiovascular or metabolic disease;
* Have history of or be diagnosed of any of the following diseases that may affect the study results: gastrointestinal disorders, hepatopathy, nephropathy, endocrine disease, blood disorders, respiratory and cardiovascular diseases;
* Currently suffering from any gastrointestinal disorders or gastrointestinal disease , including but not limited to: irritable bowel syndrome, colitis, ulcerative colitis, celiac disease, irritable bowel syndrome (IBS);
* Had hospitalizations within 3 months before screening;
* According to investigator's judgment, current frequent users of drugs may affect the gastrointestinal function or immune system.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline of gastrointestinal symptom VAS scores | Baseline (day 1 for phase 1 and day 15 for phase 2, before product consumption), at the end of the 5-day product consumption (day 5 for phase 1 and day 19 for phase 2)
  were self-measured by study subjects on a scale from 0 (never) to 3 (always) at baseline (day 1 for phase 1 and day 15 for phase 2, before product consumption) and at the end of the 5-day product consumption (day 5 for phase 1 and day 19 for phase 2).

SECONDARY OUTCOMES:
Stool frequency | Day -4, -3, -2, -1, 0, 1, 2, 3, 4, 5, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19
  In each study phase, the number of defecation per day measured during the last 5 days of wash-out period (day -4, -3, -2, -1, 0 in phase 1 and day 10, 11, 12, 13, 14 in phase 2) and the 5 days of product intervention (day 1, 2, 3, 4, 5 in phase 1 and day 15, 16, 17, 18, 19 in phase 2).
Stool consistency | Day -4, -3, -2, -1, 0, 1, 2, 3, 4, 5, 10, 11, 12, 13, 14, 5, 16, 17, 18, 19
  In each study phase, the score of stool consistency assessed using Bristol Stool Chart during the last 5 days of wash-out period (day -4, -3, -2, -1, 0 in phase 1 and day 10, 11, 12, 13, 14 in phase 2) and the 5 days of product intervention (day 1, 2, 3, 4, 5 in phase 1 and day 15, 16, 17, 18, 19 in phase 2).
Serum C-reactive protein (CRP) concentration | Day 1 before intervention (baseline), and day 5 (post-intervention)
  Only measured in phase 1
Serum Hemoglobin (HGB) concentration | Day 1 before intervention (baseline), and day 5 (post-intervention)
  Only measured in phase 1
Serum Interleukin-4 (IL-4) concentration | Day 1 before intervention (baseline), and day 5 (post-intervention)
  Only measured in phase 1
Serum Immunoglobulin G (IgG) concentration | Day 1 before intervention (baseline), and day 5 (post-intervention)
  Only measured in phase 1
Serum Immunoglobulin E (IgE) concentration | Day 1 before intervention (baseline), and day 5 (post-intervention)
  Only measured in phase 1
Serum Immunoglobulin G1 (IgG1) concentration | Day 1 before intervention (baseline), and day 5 (post-intervention)
  Only measured in phase 1
Serum Immunoglobulin G2a (IgG2a) concentration | Day 1 before intervention (baseline), and day 5 (post-intervention)
  Only measured in phase 1
Serum β-Casomorphin-7 (BCM-7) concentration | Day 1 before intervention (baseline), and day 5 (post-intervention)
  Only measured in phase 1
Serum Glutathione concentration | Day 1 before intervention (baseline), and day 5 (post-intervention)
  Only measured in phase 1
Serum calcium (Ca) concentration | Day 1 before intervention (baseline), and day 5 (post-intervention)
  Only measured in phase 1
Serum iron (Fe) concentration | Day 1 before intervention (baseline), and day 5 (post-intervention)
  Only measured in phase 1
Serum zinc (Zn) concentration | Day 1 before intervention (baseline), and day 5 (post-intervention)
  Only measured in phase 1
Fecal short chain fatty acids (SCFA) concentration | Day 1, Day 5, Day 15, Day 19
  Measured at baseline and post-intervention in each study phase
myeloperoxidase (MPO) | Day 1, Day 5, Day 15, Day 19
  Measured at baseline and post-intervention in each study phase
Subtle Cognitive Impairment Test (SCIT) | 16, 32, 48, 64, 80, 96, 112 and 128 millisecond on day 1; 16, 32, 48, 64, 80, 96, 112 and 128 millisecond on day 5; 16, 32, 48, 64, 80, 96, 112 and 128 millisecond on day 15; 16, 32, 48, 64, 80, 96, 112 and 128 millisecond on day 19
  Subject response time and error rate at stimulus exposure duration of 16, 32, 48, 64, 80, 96, 112 and 128 millisecond, as well as their head and tail means were recorded at baseline (day 1 for phase 1 and day 15 for phase 2) and the end of intervention (day 5 for phase 1 and day 19 for phase 2).

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Study Director — Sprim (Shanghai) Consulting Co., Ltd.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheng X, Li Z, Ni J, Yelland G. Effects of Conventional Milk Versus Milk Containing Only A2 beta-Casein on Digestion in Chinese Children: A Randomized Study. J Pediatr Gastroenterol Nutr. 2019 Sep;69(3):375-382. doi: 10.1097/MPG.0000000000002437. PMID 31305326